CLINICAL TRIAL: NCT00568750
Title: Dasatinib First-Line Treatment in Gastrointestinal Stromal Tumors. A Multi Center Phase II Trial
Brief Title: Dasatinib as First-Line Therapy in Treating Patients With Gastrointestinal Stromal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 56/07; SWS-SAKK-56/07; EU-20789; EUDRACT-2007-002047-24; CDR0000577496
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-01

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: gastrointestinal stromal tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Dasatinib is given orally 70 mg BID. Dasatinib will be continued until progression, unacceptable toxicity and up to 2 years (26 cycles, each cycle lasting 4 weeks).
  Other Names: Sprycel

SUMMARY:
RATIONALE: Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well dasatinib works as first-line therapy in treating patients with gastrointestinal stromal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of dasatinib as assessed by fusion PET/CT scan in patients with gastrointestinal stromal tumors.

Secondary

* To determine the efficacy and safety of dasatinib in these patients.
* To correlate the efficacy of dasatinib with KIT and PDGFR mutational status.
* To correlate the efficacy and safety of dasatinib with dasatinib drug exposure.
* To determine the efficacy of second-line treatment with another TK-inhibitor.

OUTLINE: This is a multicenter study.

Patients receive oral dasatinib twice daily on days 1-28. Treatment repeats every 28 days for 26 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastrointestinal stromal tumor (GIST)
* Measurable disease by conventional scans (CT scan or MRI) within 2 weeks prior to study registration
* Positive PET/CT scan with [^18F]-fluorodeoxyglucose uptake of the target lesions within 2 weeks prior to study registration
* No signs or history of CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Hemoglobin ≥ 90 g/L (transfusion allowed)
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* AST and/or ALT ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* No other malignancy within the past 5 years except for adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer
* No hypocalcemia (i.e., serum calcium ≤ lower limit of normal)
* No clinically significant cardiovascular disease, including any of the following:

  * Uncontrolled hypertension
  * Congestive heart failure within the past 6 months
  * QTc > 450 msec or major conduction abnormality (unless a cardiac pacemaker is present)
* No concurrent medical condition (e.g., active autoimmune disease or uncontrolled diabetes) that would impair the ability of the patient to participate in the study (at the judgment of the investigator) or that may increase the risk of toxicity, including any of the following:

  * Pleural or pericardial effusion of any grade
  * Clinically significant coagulation or platelet function disorder (e.g., known von Willebrand's disease)
  * Infection requiring intravenous antibiotics
  * Ongoing significant gastrointestinal bleeding
  * Nausea, vomiting, or malabsorption syndrome that could interfere with ingestion or absorption of oral dasatinib
* No known hypersensitivity to study drug

PRIOR CONCURRENT THERAPY:

* No prior therapy for GIST, particularly tyrosine kinase inhibitors at any time
* More than 30 days since prior participation in a clinical trial
* At least 7 days since prior and no concurrent potent CYP3A4 inhibitors, including any of the following:

  * Itraconazole, ketoconazole, miconazole, and voriconazole
  * Amprenavir, atazanavir, fosamprenavir, indinavir, nelfinavir, and ritonavir
  * Ciprofloxacin, clarithromycin, diclofenac, doxycycline, enoxacin, imatinib mesylate, isoniazid, ketamine, nefazodone, nicardipine, propofol, quinidine, and telithromycin
* At least 7 days since prior and no concurrent medications known to prolong the QT interval, including any of the following:

  * Quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, and dofetilide
  * Erythromycin and clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, and pimozide
  * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, and lidoflazine
* No concurrent IV bisphosphonates during the first 8 weeks of study treatment
* No other concurrent experimental drugs or anticancer therapy
* No concurrent drugs contraindicated for use with dasatinib, according to the dasatinib investigator's brochure

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-01-22 (Actual); Primary Completion 2012-01-18 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Response as assessed by fusion PET/CT scan according to EORTC PET Study Group criteria | at 4 weeks compared to baseline

SECONDARY OUTCOMES:
Best response as assessed by CT scan/MRI | according to RECIST criteria
Best response as assessed by fusion PET/CT scan | at 4 weeks
Clinical benefit | Clinical benefit is defined as CR, PR, or as SD lasting at least 12 weeks, determined according to RECIST
Time to progression | calculated from registration until progression or death due to tumor
Progression-free survival | calculated from registration until progression or death
Time to treatment failure | calculated from registration until premature trial treatment termination due to any reason
Overall survival | Overall survival will be calculated from registration until death or last follow-up, up to 5 years.
Adverse drug reactions according to NCI CTCAE v3.0 | Tolerability will be assessed based on the frequency and severity of Adverse Drug Reactions (ADR) coded according to NCI CTCAE v3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Montemurro, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (18):
- Biomedicum Helsinki, Helsinki, Finland
- France (4):
  - Institut Bergonie, Bordeaux
  - Hopital Edouard Herriot - Lyon, Lyon
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Universitaetsklinikum Essen, Essen, Germany
- Switzerland (12):
  - Kantonsspital Baden, Baden
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Onkozentrum - Klinik im Park, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No